CLINICAL TRIAL: NCT00407862
Title: Telmisartan vs. Losartan in Hypertensive Patients With Impaired Glucose Tolerance: A Comparison of Their Antihypertensive, Metabolic, and Vascular Effects
Brief Title: Telmisartan and Losartan in Hypertensive IGT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TCW-02-04
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Hypertension; Impaired Glucose Tolerance
Keywords: insulin resistance; beta cell function; endothelial dysfunction
MeSH Terms: conditions — Hypertension; Glucose Intolerance; Insulin Resistance | interventions — Telmisartan; Losartan

INTERVENTIONS:
Drug: Telmisartan 80 mg
Drug: Losartan 50 mg

SUMMARY:
Inhibition of RAS delays onset of diabetes in clinical studies. Preliminary evidence suggests that telmisartan may have unique metabolic properties compared to other ARB due to activation of PPARγ.

This should be tested in comparison with an ARB that is metabolically neutral in already published studies.

H0: Telmisartan is not different from Losartan with respect to metabolic and vascular effects.

H1: Telmisartan is different from Losartan with respect to metabolic and vascular effects.

DETAILED DESCRIPTION:
Background: Both, ACE-inhibitors as well as angiotensin-II-type-1 (AT1) receptor antagonists seem to reduce the development of type-II diabetes in patients with hypertension and/or high vascular risk (1-3). The major drawback of that evidence is that it derives from post-hoc analyses in studies with rather poor metabolic phenotypisation of the populations included. Additionally, all that evidence is based on measurements of fasting plasma glucose.

In subjects with impaired glucose tolerance (IGT), insulin resistance and dysfunction of pancreatic beta-cells (in variable contribution) have already established increased postprandial hyperglycemia with a consecutively increased cardiovascular risk (4, 5). In addition they have a considerable risk for future development of manifest type-II diabetes in the range of 3-6 % within a year (6, 7). In such patients prevention of diabetes may also result in cardiovascular prevention. As subjects with IGT often exhibit a more or less pronounced metabolic syndrome, hypertension is a frequently found comorbidity and vice versa IGT is frequent in hypertensive patients suggesting a possible common soil of the two diseases (8).

Given these evidences, hypertensive subjects with IGT are a very suitable target population to study metabolic and vascular effects of an angiotensin-II-type-1-receptor antagonist.

Finally, it has to be acknowledged that insulin resistance needs to be seen in the context of the proinflammatory changes of the metabolic syndrome, the endothelial dysfunction associated and the possibly central role of the adipocyte (Fig. 1). Within that context, the hypothesis was put forward that blockade of the angiotensin system might prevent type-II diabetes via effects on fat cells (9).

Rationale: The effects of different angiotensin-II-type-1-receptor antagonists on insulin sensitivity have been investigated in various studies with different, either positive (10) or negative (11, 12) results but no in-depht investigations into detailed metabolic and vascular effects have been performed.

Telmisartan is an angiotensin-II-type-1-receptor antagonist that very recently has been described to possess the specific properties of a partial activator of PPARγ (13). This effect is not found for other comparable compunds such as losartan. Genes of whom the expression is under control of that receptor are centrally involved into the pathology of the metabolic syndrome as outlined above and activation of that receptor results in improved insulin sensitivity, ameliorated endothelial dysfunction, reduced inflammation and potentially preserved beta-cell function (for review see (14)). Therefore, telmisartan is a candidate that might possess very specific beneficial properties in addition to its antihypertensive effects.

Objective: To compare the metabolic and vascular effects of telmisartan and metoprolol in hypertensive patients with IGT.

ELIGIBILITY:
Inclusion Criteria:

* IGT according the criteria of the WHO
* standardised office blood pressure > 140/90 mmHG or treated hypertension
* 40 - 75 years of age
* signed informed consent

Exclusion Criteria:

* known hypersensitivity towards telmisartan or losartan
* concommitant treatment with ACE-inhibitors
* BMI > 35 kg/m2
* inability to perform self-control of blood pressure
* acute coronary syndrome or cerebrovascular event within the last 3 months
* Revascularisation within the last 3 months
* heart failure > NYHA 2

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-01; Study Completion 2006-06

PRIMARY OUTCOMES:
HOMA index
ISI
FMD
Blood pressure surge in the morning

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Wascher, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria